CLINICAL TRIAL: NCT06689878
Title: Mobile Cognitive Behavioral Therapy for Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-04027396
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Anxiety; Stroke; Depression
Keywords: stroke recovery; stroke rehabilitation; cognitive behavioral therapy; CBT
MeSH Terms: conditions — Anxiety Disorders; Stroke; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm Using the Mobile Cognitive Behavioral Therapy App (Experimental): All participants will receive the same intervention arm, a mobile cognitive behavioral therapy (CBT) app that includes modules with educational content and teaching and practice of strategies that address the following: education about anxiety and depression and their association with stroke recovery; awareness and monitoring of emotions; behavioral activation, i.e., increasing engagement in valued and meaningful activities; increasing awareness of thinking errors and reframing negative thoughts; mindfulness; relaxation skills; increasing tolerance of anxiety in anxiety-provoking situations; and problem-solving. The application includes an interactive dashboard to provide the user with statistics for tracking progress toward their goals. Participants will be asked to use the application for 30 minutes per day, 2 days per week, for 8 weeks.
  Interventions: Behavioral: Mobile Cognitive Behavioral App

INTERVENTIONS:
Behavioral: Mobile Cognitive Behavioral App — A mobile cognitive behavioral therapy (CBT) app called "Maya" that includes modules with educational content and teaching and practice of strategies that address depression and anxiety after stroke.
  Other Names: Maya

SUMMARY:
This study aims to assess the feasibility and acceptability of "MAYA", a mobile cognitive behavioral therapy app for anxiety and mood disorders, in adults who have had a stroke.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the feasibility and acceptability of "MAYA", a mobile CBT application, in adults who have had a stroke. Feasibility will be measured by the total number of sessions completed and acceptability will be measured by scores on the Mobile Application Rating Scale-User Version (uMARS). Qualitative feedback will also be collected with a questionnaire using open-ended questions.

A secondary objective will be to evaluate preliminary efficacy of the mobile CBT application on symptoms of depression and anxiety assessed using (1) interview-based measures (the Montgomery Asberg Depression Rating Scale [MADRS] and the Hamilton Anxiety Rating Scale [HAM-A]), and (2) a patient reported outcome measure (the 21-item Depression, Anxiety, and Stress Scale [DASS]).

This study will collect pilot data over the course of 8 weeks. Because this is a pilot study, all participants will use the same version of the app and there will be no control group. Primary outcome measures will be collected at baseline (pre-intervention) and at the endpoint (week 8). Participants will be asked to use the mobile app for at least two days a week, for 30 minutes on each day, for 8 weeks. Participants will have weekly check-ins in person or via a HIPAA compliant virtual meeting platform (Zoom) with a study staff member to assess intervention adherence and answer brief questionnaires designed to assess feasibility, acceptability, and mood symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-79
* Presence of clinically-significant anxiety and/or depression (as determined by an eligibility evaluation)
* Stroke that occurred 1 month or more prior to study initiation
* Capacity to provide consent
* No greater than mild cognitive difficulties based on an eligibility evaluation conducted as part of the study
* If taking medication for depression and/or anxiety, must be on a stable dose for a minimum of 8 weeks prior to study initiation
* Ability to use iPhone or iPad independently
* Home internet access
* Willingness to participate in the full study duration.

Exclusion Criteria:

* Aphasia of moderate or greater severity (as determined during an eligibility evaluation)
* Non-fluency in English
* History of a bipolar or psychotic disorder
* Current alcohol or substance use disorder
* Active suicidal ideation
* Current engagement in psychotherapy is not grounds for exclusion unless the individual's psychotherapy is primarily focused on CBT
* Severe depression and/or anxiety based on the initial evaluation and clinical judgment of the study doctor, which warrants a higher level of care and/or immediate referral to psychiatric services
* Any other clinical or medical reason in the study doctor's initial screening evaluation that suggests the study is not appropriate for the participant

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability of MAYA as measured by the Mobile Application Rating Scale-User Version (uMARS) | Week 4 of treatment
  Feasibility and acceptability will be measured by the scores collected on the uMARS by assessing the sub scores of Engagement, Functionality, Aesthetics, and Information of the app to measure the perceived quality of the app. The outcome is the mean of the individual items, ranging from 1 to 5, with 1 denoting minimal satisfaction/rating of app quality and 5 denoting maximum satisfaction and highest rating of app quality.
Feasibility and Acceptability of MAYA as measured by the Mobile Application Rating Scale-User Version (uMARS) | Week 8 of treatment
  Feasibility and acceptability will be measured by the scores collected on the uMARS by assessing the sub scores of Engagement, Functionality, Aesthetics, and Information of the app to measure the perceived quality of the app. The outcome is the mean of the individual items, ranging from 1 to 5, with 1 denoting minimal satisfaction/rating of app quality and 5 denoting maximum satisfaction and highest rating of app quality.
Number of Sessions completed over study time period | Week 1 to Week 8 (8 week treatment)
  To assess the feasibility of "MAYA" in adults who have had a stroke, by assessing the number of sessions completed.
Qualitative Interview | Week 8 of treatment
  This is a series of questions with open-ended responses that are designed to ask participants about their experience using the app and completing the CBT program. There is no numerical scoring; responses are evaluated qualitatively to explore engagement with the app.

SECONDARY OUTCOMES:
Change in depression symptoms, as measured by the Montgomery Asberg Depression Rating Scale (MADRS) | Baseline, Week 4, and Week 8 of treatment (8 week treatment)
  Change in score on the MADRS, a clinician-rated assessment of depression symptom severity that consists of 10 items; each item is rated on a 0-6 scale, resulting in a maximum total score of 60 points, with higher scores indicative of greater depression symptom severity.
Change in anxiety symptoms, as measured by the Hamilton Anxiety Rating Scale (HAM-A) | Baseline, Week 4, and Week 8 of treatment (8 week treatment)
  Change in score on the HAM-A, a clinician-rated assessment of anxiety symptom severity that consists of 14 items; each item is rated on a 0-4 scale, resulting in a maximum total score of 56 points, with higher scores indicative of greater anxiety symptom severity.
Change in depression, anxiety, and stress, as measured by the Depression, Anxiety, and Stress Scale (DASS) | Baseline, Week 4, and Week 8 of treatment (8 week treatment)
  Change in score on the DASS, a patient-reported symptom measure of depression, anxiety, and stress symptom severity that consists of 21 items; each item is rated on a 0-3 scale, resulting in a maximum total score of 63 points, with higher scores indicative of greater depression, anxiety, and/or stress symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Jaywant, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data including demographic and clinical characteristics of individual participants as well as scores on the primary, secondary, and exploratory outcome measures.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: At the conclusion of the study, and after the researchers publish their main results, a deidentified database of individual participants will be available for data sharing. This database will be available for at least six years following the publication of the main results.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. All researchers requesting data will commit to using the data solely for research purposes; will have data shared that are pertinent to their research question/hypotheses; secure the data; return or destroy it once analyses are completed; do not share it with other researchers.

REFERENCES:
- [Background] Wilhelm S, Weingarden H, Ladis I, Braddick V, Shin J, Jacobson NC. Cognitive-Behavioral Therapy in the Digital Age: Presidential Address. Behav Ther. 2020 Jan;51(1):1-14. doi: 10.1016/j.beth.2019.08.001. Epub 2019 Aug 8. PMID 32005328
- [Background] Wang SB, Wang YY, Zhang QE, Wu SL, Ng CH, Ungvari GS, Chen L, Wang CX, Jia FJ, Xiang YT. Cognitive behavioral therapy for post-stroke depression: A meta-analysis. J Affect Disord. 2018 Aug 1;235:589-596. doi: 10.1016/j.jad.2018.04.011. Epub 2018 Apr 5. PMID 29704854
- [Background] Wada Y, Otaka Y, Yoshida T, Takekoshi K, Takenaka R, Senju Y, Maeda H, Shibata S, Kishi T, Hirano S. Effect of Post-stroke Depression on Functional Outcomes of Patients With Stroke in the Rehabilitation Ward: A Retrospective Cohort Study. Arch Rehabil Res Clin Transl. 2023 Aug 2;5(4):100287. doi: 10.1016/j.arrct.2023.100287. eCollection 2023 Dec. PMID 38163038
- [Background] Bress JN, Falk A, Schier MM, Jaywant A, Moroney E, Dargis M, Bennett SM, Scult MA, Volpp KG, Asch DA, Balachandran M, Perlis RH, Lee FS, Gunning FM. Efficacy of a Mobile App-Based Intervention for Young Adults With Anxiety Disorders: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2428372. doi: 10.1001/jamanetworkopen.2024.28372. PMID 39163044
- [Background] Mitchell AJ, Sheth B, Gill J, Yadegarfar M, Stubbs B, Yadegarfar M, Meader N. Prevalence and predictors of post-stroke mood disorders: A meta-analysis and meta-regression of depression, anxiety and adjustment disorder. Gen Hosp Psychiatry. 2017 Jul;47:48-60. doi: 10.1016/j.genhosppsych.2017.04.001. Epub 2017 Apr 3. PMID 28807138
- [Background] Ahrens J, Shao R, Blackport D, Macaluso S, Viana R, Teasell R, Mehta S. Cognitive -behavioral therapy for managing depressive and anxiety symptoms after stroke: a systematic review and meta-analysis. Top Stroke Rehabil. 2023 May;30(4):368-383. doi: 10.1080/10749357.2022.2049505. Epub 2022 Mar 30. PMID 35352629